CLINICAL TRIAL: NCT00901732
Title: Caphosol for the Reduction of Mucositis in Patients Receiving Radiation Therapy for Head and Neck Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Michael Manyak, MD / Medical Monitor, EUSA Pharma (USA), INc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 603EUSA03
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Oral Mucositis
Keywords: Caphosol; Oral Mucositis; Eusa Pharma; Moffitt Cancer Center
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Caphosol — Oral Mouth Rinse
  Other Names: supersaturated solution of calcium and phosphate ions.

SUMMARY:
Patients who have been diagnosed with a head and/or neck cancer commonly develop oral mucositis (OM). The purpose of this study is to estimate the effect of Caphosol on OM and to evaluate if Caphosol had any effect on clinical outcomes which include quality of life, oral intake, swallowing function and pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Head and Neck Cancer patients with planned Radiation therapy
* Have at least one of 10 pre-defined anatomic mucosal subsites on view
* Age >/= 18 years
* Life expectancy >/= 6 months
* Planned RT to the head/neck
* Must be able to perform oral rinse

Exclusion Criteria:

* Active infections of oral cavity
* physiologic condition that precludes the use of an oral rinse
* Hypersensitivity to Caphosol ingredients
* Presence of mucosal ulceration at baseline
* Poorly controlled hypertension, DM or other serious medical/psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to estimate ht incidence of OM in H&N cancer patients undergoing radiation therapy with or without chemotherapy and/or sensitizer who receive Caphosol. | 15 weeks

SECONDARY OUTCOMES:
The secondary objective of this study is to correlate components of OM data with clinical outcomes (pain, narcotic use, oral intake) | 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andy M Trotti, MD, Principal Investigator — Moffitt Cancer Center, Tampa Florida; David M Brizel, MD, Study Director — Duke University, Durham, North Carolina; David I Rosenthal, MD, Principal Investigator — MD Anderson Cancer Center, Houston, Texas; Mark Chambers, MD, Study Director — MD Anderson Cancer Center, Houston, Texas; Curtis T Miyamoto, MD, Study Director — Temple University Hospital, Philadelphia, PA; Kenneth Hu, MD, Study Director — Beth Israel Medical Center, New York, New York; Robert Amdur, MD, Study Director — University of Florida, Gainesville, Florida
Locations (6):
- United States (6):
  - University of Florida College of Medicine, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Beth Israel Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas